CLINICAL TRIAL: NCT01595594
Title: Effect of a PDT Protocol With Multiple Applications as an Adjuvant on the Non Surgical Treatment of Periodontal Disease in Patients With Type 2 Diabetes. A Clinical and Laboratorial Study in Humans
Brief Title: Comparison Between aPDT and Systemic Doxycycline on Non-surgical Periodontal Therapy in Type 2 Diabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Arthur Belem Novaes Jr, Chairman, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FAPESP
Record Dates: First submitted 2011-08-15; First posted 2012-05-10 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Periodontal Disease; Type 2 Diabetes
Keywords: Periodontal Diseases; Type 2 Diabetes Mellitus; hemoglobin A1c protein
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Systemic Doxycycline (Active Comparator)
  Interventions: Drug: Systemic Doxycycline and Sham aPDT
- aPDT+ Placebo (Experimental)
  Interventions: Drug: aPDT + Doxycycline Placebo

INTERVENTIONS:
Drug: Systemic Doxycycline and Sham aPDT — It will be prescribed a protocol of 100mg/day of Systemic Doxycycline for 14 days
  Other Names: aPDT Sham
  Arms: Systemic Doxycycline
Drug: aPDT + Doxycycline Placebo — The aPDT protocol will consist in 5 applications on the experimental time 0, 1, 5, 7 and 14 days.
  Arms: aPDT+ Placebo

SUMMARY:
The objective of this study is to evaluate Photodynamic Therapy (PDT) as adjunct on non surgical periodontal therapy in patients with type 2 diabetes. A total of 40 individuals will be selected and divided in two groups. On the treatment stage, the control group (Group C) will receive standard non surgical periodontal treatment. The Test Group (Group T) will be treated with PDT as an adjunct to non surgical periodontal treatment. The treatment will be repeated 4 times in two weeks, followed by dental prophylaxis every 15 days until accomplish 3 months. The follow-up will be done for 6 months. The clinical parameters measured will be: plaque index, pocket depth, bleeding on probing, relative clinical insertion level and suppuration. In addition, the evaluation of crevicular fluid volume and the levels of IL-1, TNF-α, subgingival microbiota by the hybridization DNA-DNA Checkerboard technique. The investigators expect to find identical or better results for the test group.

ELIGIBILITY:
Inclusion Criteria:

* Poorly Controlled Type 2 Diabetes (HbA1c > 7%)
* Advanced Chronic Periodontitis
* Presence of 15 teeth

Exclusion Criteria:

* Use on antiinflammatory drugs
* Use of antibiotics less then 6 months before therapy
* Smokers
* Positive for HIV
* Periodontal treatment less then 6 months before therapy
* Advanced complications of Diabetes

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level | 0, 1 month, 3 months and 6 months
  There will be analyzed the changes in clinical attachment level at the proposed experimental times. Clinical attatchment level is known as a proper outcome to evaluate periodontal disease progression or regression. It is measured as the distace between the deepet point fo the periodontal pocket and a stabilshed point, on the case of this study, the tooth occlusal surface.

SECONDARY OUTCOMES:
Microbial Load | 0, 3 months and 6 months
  There will be mesaured the changes of microbial load at the proposed experimental times. Microbial load at deep pocket seems to change regarding periodontal treatment and it is expected a reduction after treatment. measuring on various experimental times it will be possible to evaluate treatment stability on reducing periodontopathogens.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Odontologia de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Result] O'Connell PA, Taba M, Nomizo A, Foss Freitas MC, Suaid FA, Uyemura SA, Trevisan GL, Novaes AB, Souza SL, Palioto DB, Grisi MF. Effects of periodontal therapy on glycemic control and inflammatory markers. J Periodontol. 2008 May;79(5):774-83. doi: 10.1902/jop.2008.070250. PMID 18454655
- [Result] Lulic M, Leiggener Gorog I, Salvi GE, Ramseier CA, Mattheos N, Lang NP. One-year outcomes of repeated adjunctive photodynamic therapy during periodontal maintenance: a proof-of-principle randomized-controlled clinical trial. J Clin Periodontol. 2009 Aug;36(8):661-6. doi: 10.1111/j.1600-051X.2009.01432.x. Epub 2009 Jun 25. PMID 19563331
- [Derived] Ramos UD, Ayub LG, Reino DM, Grisi MF, Taba M Jr, Souza SL, Palioto DB, Novaes AB Jr. Antimicrobial photodynamic therapy as an alternative to systemic antibiotics: results from a double-blind, randomized, placebo-controlled, clinical study on type 2 diabetics. J Clin Periodontol. 2016 Feb;43(2):147-55. doi: 10.1111/jcpe.12498. Epub 2016 Feb 19. PMID 26710892